CLINICAL TRIAL: NCT03743376
Title: The HIV Functional Cure Potential of UB-421: A Phase II, Randomized, Open-label, Controlled, 48 Week, Proof of Concept Study, to Evaluate the Safety of UB-421 in Combination With Standard Antiretroviral Therapy (ART) and the Efficacy of HIV Reservoir Reduction as Compared With ART Alone in ART Stabilized HIV-1 Patients
Brief Title: The HIV Functional Cure Potential of UB-421 in ART Stabilized HIV-1 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United BioPharma (Industry)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Taoyuan General Hospital (Other Government); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A209-HIV
Record Dates: First submitted 2018-11-12; First posted 2018-11-16 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — UB-421

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard ART (No Intervention): Subjects will receive standard ART for 48 weeks
- UB-421(25mg/kg) Q2W add-on treatment (Experimental): UB-421(25 mg/kg) Q2W plus standard ART for 48 weeks
  Interventions: Biological: UB-421(25 mg/kg) Q2W
- UB-421(25mg/kg) Q4W add-on treatment (Experimental): UB-421(25 mg/kg) Q4W plus standard ART for 48 weeks
  Interventions: Biological: UB-421(25 mg/kg) Q4W

INTERVENTIONS:
Biological: UB-421(25 mg/kg) Q2W — Monoclonal antibody by IV infusion plus standard ART
  Arms: UB-421(25mg/kg) Q2W add-on treatment
Biological: UB-421(25 mg/kg) Q4W — Monoclonal antibody by IV infusion plus standard ART
  Arms: UB-421(25mg/kg) Q4W add-on treatment

SUMMARY:
This study evaluate the safety of UB-421 in combination with standard antiretroviral therapy (ART) and the efficacy of HIV reservoir reduction as compared with ART alone in ART stabilized HIV-1 patients

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 sero-positive
2. Male with body weight ≥ 50 kg or female with body weight ≥ 45 kg.
3. HIV-1 plasma RNA level below 50 RNA copies/mL .

Exclusion Criteria:

1. Subjects with active systemic infections, except for HIV-1, that the Investigator feels the infections may confound evaluation and treatment for HIV-1.
2. Current active hepatitis B carriers, ie, hepatitis B surface antigen positive.
3. Current active hepatitis C carriers, ie, hepatitis C virus (HCV) antibody positive.
4. History of anaphylaxis to other mAbs.
5. Any vaccination within 8 weeks prior to the first dose of assigned drug.
6. Use of immunomodulators, HIV vaccine, or systemic chemotherapy within 180 days prior to the first dose of assigned drug.
7. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
treatment related TEAEs | 48Weeks
  the incidence of Grade 3 drug-related treatment-emergent adverse events

SECONDARY OUTCOMES:
the change of immune profiles | 16Weeks
  Change in Treg percentage in the peripheral blood

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei